CLINICAL TRIAL: NCT01133743
Title: An Open-Label Phase 2 Study of Lenalidomide (Revlimid) in Combination With Oral Dexamethasone in the Treatment of Previously Untreated, Symptomatic Patients With Chronic Lymphocytic Leukemia (CLL)
Brief Title: Open-Label Study of Lenalidomide in Combination With Oral Dexamethasone in the Treatment of Previously Untreated, Symptomatic Patients With Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RV-CLL-PI-0411
Record Dates: First submitted 2010-05-19; First posted 2010-05-31 (Estimated); Last update posted 2017-05-03 (Actual); Status verified 2017-05

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: Lenalidomide; Dexamethasone; Immunomodulatory Drugs(IMiD™); Thalidomide analogues
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Lenalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lenalidomide and Dexamethasone (Experimental): Lenalidomide target dose of 25 mg PO OD continuously (28-day cycle) using an initial dose escalation period. Oral dexamethasone 12 mg daily on days 1-7, 14 and 21 of each cycle.
  Interventions: Drug: Lenalidomide and Dexamethasone

INTERVENTIONS:
Drug: Lenalidomide and Dexamethasone — Starting Lenalidomide dose 2.5 mgs or 5 mgs (based on baseline calculated creatinine clearance)PO daily on a 28 day cycle. Dose escalations will take place at the start of subsequent cycles as frequently as tolerated but not more frequently than at the start of each cycle to a target dose of 25mg daily. Oral dexamethasone at 12 mg PO daily will be administered on days 1-7, 14 and 21 of each cycle
  Other Names: Lenalidomide; Immunomodulatory drug(IMiD™); Thalidomide analogues

SUMMARY:
This is a phase II, non-randomized, single institution study in symptomatic, previously untreated CLL patients. All patients will receive the study drug, lenalidomide, given PO daily continuously on a 28 day cycle at the starting dose level of either 2.5 mgs or 5 mgs with dose escalations to a target dose of 25mg daily. Oral dexamethasone at 12 mg PO daily will be administered on days 1-7, 14 and 21 of each cycle. Patients will be treated with lenalidomide and dexamethasone to 2 cycles past CR or to a maximum of 18 cycles, each cycle of 28 days duration. Primary endpoint is response.

ELIGIBILITY:
Inclusion Criteria

1. Understand and voluntarily sign an informed consent form.
2. Age >/=18 years at the time of signing the informed consent form.
3. Able to adhere to the study visit schedule and other protocol requirements.
4. A confirmed diagnosis of B-cell CLL by IWCLL 2008 criteria
5. No prior systemic therapy for CLL. Steroid therapy alone for autoimmune cytopenias (anemia or thrombocytopenia) is NOT considered a prior systemic therapy.

   Radiation: Patients may have received prior radiation therapy restricted to </= 25% of functioning bone marrow. Patients must be >/= 4 weeks since last treatment with radiation therapy.

   Surgery: previous surgery is permissible. Patient must be >/= 4 weeks since any major surgery.
6. Patients must have symptomatic disease requiring therapy as per the IWCLL 2008 criteria. One or more of the following must be present to be eligible:

   * Massive (>10cm diameter), progressive or symptomatic lymphadenopathy
   * Massive (>6 cm below costal margin) or progressive or symptomatic splenomegaly
   * Anemia (Hb <110 g/L)
   * Thrombocytopenia (platelets <100 x 109/L)
   * Constitutional symptoms (one of the following):
   * Weight loss >10% or more over previous 6 months
   * Significant fatigue
   * Fevers >38 degrees Celsius for 2 or more weeks without infection
   * Night sweats > 1 month without evidence of infection
   * Other constitutional symptoms felt to require treatment as per treating physician discretion
   * Persistent rise in lymphocyte count with doubling time of < 6 months
   * Autoimmune anemia and/or thrombocytopenia poorly responsive to corticosteroids or other standard therapy
7. ECOG performance status of </= 2 at study entry
8. Laboratory Requirements: (must be done within 7 days prior to first study drug dose) Hematology: Absolute granulocytes (AGC)>/= 1000/mm³ Platelets >/= 50,000/mm³ Chemistry: Creatinine clearance>/= 30ml/min (by Cockcroft-Gault calculation, see Appendix 9) Bilirubin </= 1.5 x UNL AST (or ALT if AST not available) </= 2.5 x UNL
9. Females of childbearing potential (FCBP)† must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL within 10 - 14 days prior to and again within 24 hours of starting lenalidomide and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking lenalidomide. FCBP must also agree to ongoing pregnancy testing. Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy. All patients must be counseled at a minimum of every 28 days about pregnancy precautions and risks of fetal exposure.
10. Disease free of prior malignancies for >/= 5 years with exception of currently treated basal cell, squamous cell carcinoma of the skin, or carcinoma "insitu" of the cervix or breast
11. Able to take aspirin 81 mg daily as prophylactic anticoagulation (patients intolerant to ASA may use warfarin or low molecular weight heparin).

Exclusion criteria:

Patients who fulfill any of the following criteria are not eligible for admission to the study:

1. Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.
2. Pregnant or breast feeding females. (Lactating females must agree not to breast feed while taking lenalidomide).
3. Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
4. Evidence of laboratory TLS by Cairo-Bishop Definition of Tumor Lysis Syndrome. Subjects may be enrolled upon correction of electrolyte abnormalities.
5. Use of any other experimental drug or therapy within 28 days of baseline.
6. Known hypersensitivity to thalidomide.
7. The development of erythema nodosum if characterized by a desquamating rash while taking thalidomide or similar drugs.
8. Any prior use of lenalidomide.
9. Concurrent use of other anti-cancer agents or treatments.
10. Known positive for HIV or infectious hepatitis, type B or C.
11. Known intolerance to steroids (i.e. poorly controllable hyperglycemia or hypertension, significant mood disturbances, steroid-related myopathy, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2010-05; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Response rate | 18 cycles (each cycle is of 28 days)

SECONDARY OUTCOMES:
Time to progression | Participants will be followed until death

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Christine I Chen, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network - Princess Margaret Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Chen CI, Paul H, Snitzler S, Kakar S, Le LW, Wei EN, Lau A, Johnston JB, Gibson SB, Queau M, Spaner D, Croucher D, Sherry B, Trudel S. A phase 2 study of lenalidomide and dexamethasone in previously untreated patients with chronic lymphocytic leukemia (CLL). Leuk Lymphoma. 2019 Apr;60(4):980-989. doi: 10.1080/10428194.2018.1508669. Epub 2018 Oct 2. PMID 30277089